CLINICAL TRIAL: NCT00982761
Title: Analysis of Health Status of Occupational Driver
Brief Title: Metabolic Syndrome of Occupational Drivers
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Research Ethics Review Committee
Other Study IDs: 098012-3
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-09

CONDITIONS: Metabolic Syndrome
Keywords: occupational drivers; health status
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to discover the health status of occupational drivers. The health status includes data collection of body mass index, blood pressure, central obesity, anxiety scale scores, smoking habit and related cessation therapy, etc.

DETAILED DESCRIPTION:
Occupational drivers' health is essential for passengers' safety. However, occupational drivers' health is damaged by long-term sitting and driving, lack of exercise, stress from traffic, and irregular diet. The objectives of this study were to assess the health status of occupational drivers in Taiwan. The measures included blood pressure, central obesity, fasting blood sugar, triglyceride, body mass index (BMI), anxiety scale scores, and metabolic syndrome, etc.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome
* hypertension
* anxiety scale scores

Exclusion Criteria:

* hyperuricemia

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study is to understand the health status of occupational status. Occupational drivers work in a sitting position for long durations, facing traffic stress, irregular mealtimes and lack of exercise etc, and may impede their health. For passengers, their safety is related to the occupational drivers' health status and should pay attention to the health condition of the occupational drivers.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Yin Wu, MD, Study Chair — Chung Yin Wu